CLINICAL TRIAL: NCT05991973
Title: A Phase ll, Multi-center, Single-arm Clinical Study of Low-dose Chidamide Maintenance Therapy After Allogeneic Hematopoietic Stem Cell Transplantation for T-cell Acute Lymphoblastic Leukemia or T-cell Lymphomas
Brief Title: Low-dose Chidamide Maintenance Therapy After Allo-HSCT for T-cell Acute Lymphoblastic Leukemia or T-cell Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); The Affiliated Hospital of Medical College, Ningbo University (Other)
Responsible Party: Principal Investigator, He Huang, The President of The First Affiliated Hospital, College of Medicine, Zhejiang University, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IIT20230004C-R2
Record Dates: First submitted 2023-07-23; First posted 2023-08-15 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2024-08

CONDITIONS: T Lymphoblastic Leukemia/Lymphoma
Keywords: chidamide; allo-HSCT; maintenance therapy
MeSH Terms: conditions — Lymphoma | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- low-dose chidamide maintenance therapy after allo-HSCT (Experimental)
  Interventions: Drug: Chidamide

INTERVENTIONS:
Drug: Chidamide — Chidamide was initiated between days +30 and +100 post-transplant at 10 mg twice weekly (BIW), continued for up to 2 years (24 courses, 4 weeks as a course) or until relapse, intolerable toxicity, or withdrawal. The dose could be escalated to a maximum of 20 mg BIW if MRD became positive during treatment. Donor lymphocyte infusion (DLI) was permitted in cases of MRD positivity.

SUMMARY:
Clinical Study on the Safety and Effectiveness of low-dose chidamide maintenance therapy after allogeneic hematopoietic stem cell transplantation for T-cell acute lymphoblastic leukemia or T-cell lymphomas.

DETAILED DESCRIPTION:
This is a phase ll, multi-center, single-arm clinical study.This study is indicated for high-risk of T-cell acute lymphoblastic leukemia or T-cell lymphomas patients. It aims to evaluate the safety and effectiveness of low-dose chidamide maintenance therapy after allogeneic hematopoietic stem cell transplantation for T-cell acute lymphoblastic leukemia or T-cell lymphomas to prevent relapse. 44 patients will be enrolled. The clinical end points include relapse-free survival, acute or chronic GVHD, non-relapse mortality, and overall survival, etc.

ELIGIBILITY:
Inclusion Criteria:

1. T-cell acute lymphoblastic leukemia or T-cell lymphomas (mainly including peripheral T-cell lymphoma, NK/T-cell lymphoma, T-lymphoblastic lymphoma, etc.) must be diagnosed before enrollment. The diagnostic criteria refer to the 2016 WHO classification. Patients is in high-risk group or standard-risk group with MRD-positive patients after transplantation.
2. Age 14-70;
3. Stable hematopoietic reconstitution after receiving allogeneic hematopoietic stem cell transplantation, no aGVHD or stable aGVHD control and stable primary disease;
4. Complete donor chimerism after transplantation;
5. During the screening period after transplantation (within 4 weeks before Chidanilide administration), the primary disease is remission and MRD is negative.
6. Eastern Cooperative Oncology Group (ECOG) physical condition score is 0-2 points;
7. Creatinine clearance ≥ 60 mL/min (according to the Cockcroft-Gault formula);
8. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal range (ULN), total bilirubin ≤ 2 × ULN;
9. Echocardiography (ECHO) shows left ventricular ejection fraction (LVEF) ≥ 50%
10. Life expectancy >8 weeks;
11. Voluntarily sign the informed consent form, understand and comply with the requirements of the research.

Exclusion Criteria:

1. Bone marrow recurrence or extramedullary recurrence after transplantation;
2. Hemocytopenia after transplantation: white blood cells <2000/ul, platelets <25000/ul;
3. Active grade 3-4 acute GVHD, or active moderate-to-severe chronic GVHD that cannot be controlled by drugs;
4. Active autoimmune diseases, such as SLE, rheumatoid arthritis, etc.;
5. Currently suffering from clinically significant active cardiovascular disease, such as uncontrolled arrhythmia, prolonged QTc interval of electrocardiogram, uncontrolled uncontrolled hypertension, congestive heart failure, any New York Heart Association (NYHA) functional class 3 or 4 cardiac disease, or a history of myocardial infarction within 6 months before screening;
6. Other serious diseases that may limit patients to participate in this trial (such as advanced infection, uncontrolled diabetes, renal failure);
7. Known human immunodeficiency virus (HIV) infection, or hepatitis B virus that cannot be controlled by drugs (HBV-DNA positive, and HBV DNA test value above the upper limit of normal value) or hepatitis C virus (anti-HCV positive, and HCV viral titer detection value above the upper limit of normal value) Chronic Infect;
8. Pregnant or lactating women;
9. Those who cannot understand and follow the research protocol or cannot sign the informed consent form;

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Relapse-free survival(RFS) | At Year 2
  The time from the date of treatment to the occurrence of any of the following:
  1. Death from any cause
  2. Disease recurrence, defined as one of the following:
  Leukemia blasts reappeared in peripheral blood, or blasts ≥ 5%, naive monocytes ≥ 5% in bone marrow, or extramedullary lesions.

SECONDARY OUTCOMES:
Graft-versus-host disease (GVHD) | At Year 2
  Acute GVHD or chronic GVHD incidence after chidamide maintenance therapy
Adverse effects | At Year 2
  Drug related adverse effects after chidamide maintenance therapy
Measurable residual disease(MRD) status | At Year 2
Changes in t lymphocyte subsets | At Year 2
Non-relapse mortality (NRM) | At Year 2
  Assessment of NRM at Year 2
GVHD-free-relapse-free survival(GRFS) | At Year 2
  Assessment of GRFS at Year 2
Overall survival (OS) | At Year 2
  Assessment of OS at Year 2

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Zhejiang Medical Colleage Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No